CLINICAL TRIAL: NCT06332066
Title: Oxytocin Administration to Therapists and Its Effects on Patient-perceived Attunement and Responsiveness
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 0046-24-COM
Record Dates: First submitted 2024-03-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Mental Health Therapists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): 24IU (12IU*2) of Oxytocin, Sorbitol, Benzyl, alcohol glycerol, distilled water.
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): 24IU (12IU*2) of Sorbitol, Benzyl, alcohol glycerol, distilled water.
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal OT will be performed using a spray containing 24IU (12IU administered to each nostril), sorbitol, benzyl, alcohol glycerol, distilled water. Dosage and administration method was determined by standard OT studies instructions and guidelines. The substance will be prepared immediately after randomization by an external preparation and delivered and stored until administration under required conditions. The nasal spray will be self administered, with nursing staff supervising for proper administration of substance, and for supervision of side effects.

SUMMARY:
In recent years there is a great interest in the possible role of Oxytocin (OT) as a facilitator for enhancing psychotherapeutic processes in patients with mental illnesses. Specific studies explored OT administration to patients, and the effect on psychotherapy on interaction within the therapeutic dyad. Nonetheless, studies exploring OT's effects of the therapists' side of the therapeutic dyad on the psychotherapy session and outcome, have not been conducted. The current study aims to assess the effect of OT administration to the therapists of psychiatric outpatients, on treatment process and outcome and specifically on the patient and therapist experience of the attunement and responsiveness toward the patient in the therapeutic encounter. Twenty staff members from Teradion Mental health Clinic of Clalit Health Services will be recruited, as well as 100 patients treated by these staff members. Therapists agreeing to participate will receive OT and PLC in a random order, at the same day they are seeing the same patients and the consecutive week. Patients agreeing to participate will complete a demographic questionnaire and all study measures, and will be scheduled to perform two consecutive research sessions with their therapists. The therapist will receive either OT or PLC in each of these two sessions, and right after the session the patients will complete the assessment scales. Multilevel models will be performed by the investigators to assess the effects of OT administration in therapists receiving OT versus receiving placebo. This research will be performed in accordance with ethical principles of Helsinki WMA Declaration. This study is the first to assess the effectiveness of hormonal augmentation for therapists and its influence on therapeutic process with patients suffering from acute distress in the public mental health domain.

DETAILED DESCRIPTION:
In the past few decades, efforts have been made to explore the potential augmenting effect of neurobiological compounds for patients with mental disorders (Hertenstein et al, 2021). One of these compounds is Oxytocin (OT), a nine-amino acid neuropeptide generated in the hypothalamus and released by the pituitary gland (Brownstein et al., 1980). Oxytocin has been suggested to be one of these possible facilitators when administered in clinical settings (Peled-Avron et al., 2020). Studies show that OT administration can enhance social abilities of children with autism spectrum disorder (Yatawara et al.,, 2016; Parker et al., 2017), decrease depression and anxiety symptoms when administered as add-on to antidepressants (Scantamburlo et al., 2015), reduce anxiety and negative self-appraisal following exposure therapy (Guastella et al., 2009; Alvares et al., 2012) and improve theory of mind among patients with schizophrenia (De Coster et al., 2019; Pedersen et al., 2011; Modabbernia et al., 2013).

Aside from its potential direct neural effects, OT was previously suggested to enhance treatment outcomes through its effects on vital interpersonal processes taking place during psychotherapy. As early as 2010, OT was suggested to affect the therapeutic process through its ability to modulate trust and sense of safety, which seem crucial for effective therapeutic processes to take place (Olff et al., 2010). Indeed, studies have documented that OT administration can improve trust and cooperation in humans (Barraza & Zak, 2009; De Dreu, 2012; Xu et al, 2019). Nonetheless, in a recent study conducted by Grossman-Giron et al. (2021), OT administration led to more favorable therapeutic outcomes, but led to no improvement in the therapeutic working alliance between patients and therapists.

One biobehavioral model which can explain the compelling evidence found in Grossman-Giron et al. (2021) is the putative role of OT in the activation of the caregiving system of the therapist. Studies demonstrate that activation of the caregiving system in response to the other's distress is mediated by release of OT (Swain et al., 2012). Studies assessing the neurobiological mechanisms associating OT with caregiving behavior demonstrate that a crying infant increases activation in insula and inferior frontal gyrus in the mothers' brain, and reduces activation in right amygdala, all regions known to be involved in empathy and empathic caregiving responses (Naber et al., 2010; Riem et al., 2011; Swain et al., 2012). Similarly, elevated OT levels in the mother were found to be associated with mothers' response to their infants' stress, a trend which was evident also among foster mothers (Bick & Dozier, 2013). OT administration to fathers was also found increased parental behaviors in father-child dyads (Weisman et al., 2012). These combined findings suggest that OT's effect of vital elements of the therapeutic dyad, such as responsiveness to patients' distress and the ability to convey support, empathy, and trust, might be situated in the therapist.

Although no study has previously tested the effect of OT administration to therapist on therapeutic process and outcome, several correlative studies have provided partial support for such an effect. In a recent study conducted by Fisher et al. (2023), the authors examined therapists' hormonal response as a possible biomarker of effective therapeutic interventions. In this study, therapists' (n=6) OT levels were measured during the ongoing therapy of men (n=62) suffering from depression. The authors found that therapists' OT levels mediated the association between patients' negative emotions and depression severity. Put differently, the authors found that patients' negative emotions were associated with increased levels of OT, which in turn was associated with therapeutic outcomes. These findings might suggest that the elevation in OT system might have produced a shift in specific caregiving mechanisms which produced a more favorable outcome.

Several potential therapist-specific mechanisms might be associated with this elevation of OT occurring during psychotherapy. OT is strongly linked to empathy, which is considered a vital element of the therapeutic process (Elliott et al., 2011). Client-perceived empathy was found to be a predictor of outcome of psychotherapy (Barrett-Lennard, 1981; Elliott et al., 2011). Another potential factor likely to be associated with OT and the caregiving system is therapists' behavioral responsiveness, defined as the therapist's ability to adjust their responses to the current state of the client (Falkenstrom, 2015). In a study conducted by Wu and Levitt (2020), therapist behavioral responsiveness was assessed in a metanalysis of 75 studies. The authors found that specific responses are important in different therapeutic contexts, within psychotherapy interventions and with patients with different characteristics. Finally, it can also be speculated that activation of the caregiving system would lead to changes in attunement, defined as a process of communion and unity of interpersonal contact, going beyond empathy, to create a two-person experience of connectedness by providing a reciprocal affect and/or resonating response (Erskine, 1998). Studies demonstrate that the higher the attunement, the better the outcome (Aafjes-van Doorn et al. 2022). Taken together, these three therapist-specific factors, and how they are specifically perceived by the patient, might be stronger mediators between OT and therapy outcomes.

To the best of our knowledge, no study has thus far examined whether OT augmentation to therapists might affect their therapeutic response, as perceived by their patients. This study aims to bridge this gap in scientific knowledge by testing the effect of OT administration to therapists on patient-perceived therapist empathy, therapist behavioral responsiveness and therapists' attunement. Finally, we aim to explore the mediational effect of these constructs on changes in patients' distress.

Study Hypotheses

1. Patients in the IN-OT sessions will experience the therapist as more empathic, attuned and responsive, as opposed to the placebo encounter.
2. Levels of distress in the session after OT administration will be lower compared to the levels of distress in the session after PLC administration.
3. Perceived empathy, responsiveness and attunement will mediate the association between OT administration and patient distress.

Methods Participants Twenty staff members from Teradion Mental health Clinic of Clalit Health Services will be recruited, as well as 100 patients treated by these staff members. Inclusion criteria for therapists will be: psychotherapists in different stages of professional training, in adult clinic, who meet patients for individual therapy. Exclusion criteria for therapists will be psychotherapists self-declaring pregnancy or breastfeeding. Inclusion Criteria for patients will be: patients coming for regular therapy once or twice a week. Exclusion Criteria for patients will be: an inability for any reason to complete self-report questionnaire, or terminating treatment between study trials.

Measures Process measures The Patient's Experience of Attunement and Responsiveness Scale (PEAR; Snyder & Silberschatz, 2017). A self-report measure designed to assess the patient's experience of the therapist's degree of attunement and responsiveness during a therapy session. The items that comprise the scales are based on clients rating their therapy experiences overall at the end of the treatment meeting, and therapists rating the same scales, separately (Silberschatz, 2012; Silberschatz, Curtis, Sampson, & Weiss, 1991). For the purpose of the current study, only the patient version will be utilized. The PEAR patient version (PEAR-p) contains 20 statements, pertaining to attunement and responsiveness for example: "My therapist had accurate empathy for my needs and feelings today", "What my therapist did and said was helpful today". Participants rate each item on a Likert scale that ranges from 0 to 3, which are then summed to achieve a total attunement and responsiveness score. Patient's experience of attunement and responsiveness may be comprised of three distinct factors that assess the patient's perceptions of: (1) the therapist's helpful actions during a session,(2) the therapist's empathy and caring during a session, and (3) the patient's sensed accomplishments during a therapy session. The Patient version of the PEARS demonstrated good reliability with coefficient ω =.94 as did the Therapist version with coefficient ω=.96 Attachment Formation (AF; Fraley & Davis, 1997). The AF is a six-item self-reported measure assessing attachment-related functions. The AF closely follows the theoretical model proposed by Bowlby (1969, 1977, 1982), and is based on the three functions an attachment figure should fulfill based on attachment theory: proximity seeking, safe haven, and secure base. Items were rated on a 5-point Likert scale ranging from 1 (Disagree) to 5 (Strongly agree). In the current study, we adapted this measure to examine the development of attachment formation to the therapist, to assess the extent to which the therapist serves as an attachment figure. Internal consistency for attachment formation was .77. The Pear will be completed by patients after each encounter.

The Working Alliance Inventory - Short Revised (WAI - SR; Hatcher & Gillapsy, 2006). A 12-item self-report questionnaire aimed to evaluate patient-therapist working alliance through three aspects: agreement on therapy goals, agreement on therapeutic tasks and patient-therapist positive emotional bond. The WAI-SR is a brief version of the original 36-item WAI (Horvath & Greenberg, 1989), and an extended version of the 6-item Working Alliance Inventory (WAI-6; Falkenström et al., 2014). It is rated on a 6-point scale ranging from not at all (1) to very much (6). The questionnaire has two versions: one assessing the alliance from the patient's point of view (see Appendix C) and the other assessing it from the therapist's point of view (see Appendix D). It was translated to Hebrew by Milhade (2018). The WAI-SR has demonstrated excellent reliability, convergent validity, and predictive validity (MacFarlane et al., 2015). Patients will complete the WAI-12 after each encounter.

Outcome Measures The Hopkins symptoms checklist -short form (HSCL-11; Lutz, Tholen, Schürch, & Berking, 2006). The HSCL-11 is a brief version of the SCL-90-R (Derogatis et al., 1992) and includes 11 items assessing general symptomatic distress through self-report (see Appendix A). The HSCL-11 is highly correlated with the Global Severity Index (r = .91) and has high internal consistency (Lutz et al., 2006). The HSCL-11 was previously found suitable for detecting weekly changes in symptom severity during the course of treatment in major depression disorder patients (Lutz, Stulz, & Köck, 2009). In order to assess changes in general distress, as manifested by anxiety and depression symptoms. The HSCL-11 will be delivered after the therapeutic encounter.

Procedure Therapists agreeing to participate will receive OT and PLC in a random order, at the same day they are seeing the same patients and the consecutive week (to illustrate, therapist 1 can be randomly assigned to receive OT on Monday, and PLC the next Monday, when the same patients will arrive to the clinic). The clinic nurse will be handling inhalers and will also be blind to content (OT vs. placebo). Patients agreeing to participate will complete a demographic questionnaire and all study measures (this will be considered as baseline measurement), and will be scheduled to perform two consecutive research sessions with their therapists. The therapist will receive either OT or PLC in each of these two sessions, and right after the session the patients will complete the assessment scales.

Dosing Human (IN-OT) studies primarily employ dosages between 20 and 48 IU )Grace et al., 2018), with the majority using a 24 IU dose. OT administration benefits as treatment add-on were shown to be influenced by dose magnitude (Yamasue et al., 2022; Le et al., 2022). This study will therefore use 24IU inhalers lasting for 07 hours, allowing therapist to see 4-5 patients on the day of research participation.

Statistical strategy Multilevel models (MLM, Bosker & Snijders, 2011) will be performed by the investigators to assess the effects of OT administration in therapists receiving OT versus receiving placebo. The Preacher and Hayes (2008) approach will be employed for the purposes of assessing the mediating role of responsiveness, attunement and empathy on the association between OT administration and outcome. Statistical analyses will be performed using the Statistical Package for the Social Sciences (SPSS) v.25 (IBM Corp. Armonk, NY, USA) as well as in R Version 4.1.0 package 'nlme' (Pinheiro, Bates, DebRoy, & Sarkar, 2016).

Ethical considerations This research will be performed in accordance with ethical principles of Helsinki WMA Declaration. As such, the rights, safety and welfare of the study's participants will be prioritized. Therapists and patients will sign informed consent forms before participating in any study related procedures. Participants will be able to leave the study at any time and they will be informed that leaving the study will not affect their work or treatment. The current study is submitted for the approval of the Institutional Review Board (IRB) committee of Shalvata Mental Health Center.

Information safety Clinical data obtained from the facilities of Teradion MHC, and the participants' blinded data will be collected and stored on safely guarded computers of Clalit Health Services. Data will be completely anonymized.

Importance and novelty of the proposed study This study is the first to assess the effectiveness of hormonal augmentation for therapists and its influence on therapeutic process with patients suffering from acute distress in the public mental health domain. Previous studies exploring the effect of OT have applied OT as an add on to treatment, by giving it directly to the patient, and have shown different outcomes on patients' improvement. Furthermore, the study will provide important insights related to the mediating influence of OT on her attunement and responsiveness to the patient.

ELIGIBILITY:
Inclusion Criteria for Therapists:

Psychotherapist (psychologists, psychiatrists, social workers, dieticians, and art therapists in different stages of seniority and training) in adult clinic and eating disorder clinic , who encounter patients for individual therapy will be included.

Exclusion Criteria for Therapists:

Psychotherapists self-declaring pregnancy or breastfeeding.

Inclusion Criteria for Patients:

Patients coming for regular therapy once or twice a week

Exclusion Criteria for Patients:

Patients leaving treatment at time of trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Attunement and Responsiveness towards patients | 3 weeks
  PEAR; Snyder & Silberschatz, 2017 - The Patient's Experience of Attunement and Responsiveness Scale

SECONDARY OUTCOMES:
Attachment with Therapist | 3 weeks
  AF; Fraley & Davis, 1997 - Attachment Formation toward the therapist
Working Alliance with Therapist | 3 weeks
  The Working Alliance Inventory - Short Revised (WAI - SR; Hatcher & Gillapsy, 2006).
Patient Symptoms | 3 weeks
  The Hopkins symptoms checklist -short form (HSCL-11; Lutz, Tholen, Schürch, & Berking, 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Clinic, Teradion, Misgav Regional Council, Israel